CLINICAL TRIAL: NCT02994953
Title: A Phase Ib Open-Label, Dose-Finding Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Avelumab in Combination With M9241(NHS-IL12) in Subjects With Locally Advanced, Unresectable, or Metastatic Solid Tumors
Brief Title: A Phase Ib Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) of Avelumab in Combination With M9241(NHS-IL12) (JAVELIN IL-12)
Acronym: COMBO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to pre-specified futility criteria met.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201781_0031; 2017-002212-13 (EudraCT Number)
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors
Keywords: Avelumab; M9241; NHS-IL12; Advanced Solid Tumors
MeSH Terms: interventions — avelumab; Maximum Tolerated Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 4 micrograms per kilogram (mcg/kg) a subcutaneous (SC) injection at time (up to -20 minutes) relative to the start of Avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks on Day 1 and 15 during each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
  Interventions: Drug: Avelumab; Drug: M9241; Drug: M9241 (MTD)
- Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
  Interventions: Drug: Avelumab; Drug: M9241
- Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 12 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
  Interventions: Drug: Avelumab; Drug: M9241
- Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
  Interventions: Drug: Avelumab; Drug: M9241
- Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg (Experimental): Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 800 milligrams (mg) IV infusion once weekly for the first 12 weeks, then 800 mg once every 2 weeks of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
  Interventions: Drug: Avelumab (Once weekly)
- Part B Cohort 1: UC Cohort Stage 1 combination therapy (Experimental): Participants in the expansion cohorts received M9241 at dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks on Day 1 in combination with Avelumab 800 mg IV infusion once weekly for the first 12 weeks, then 800 mg once every 2 weeks of each cycle (Each cycle=28 days) determined as the RP2D in the escalation part of the study.
  Interventions: Drug: Avelumab (Once weekly); Drug: Avelumab (Expansion cohort)

INTERVENTIONS:
Drug: Avelumab — Participants received avelumab intravenous (IV) infusion once a week on Day 1 and Day 15 of each cycle.
  Other Names: MSB0010718C
  Arms: Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg
Drug: M9241 — Participants received Subcutaneous (SC) injection of M9241 in escalating doses on Day 1 of each cycle.
  Arms: Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg
Drug: Avelumab (Once weekly) — Participants received avelumab once weekly in combination with M9241 every 4 weeks at M9241 maximum tolerated dose (MTD) for first 12 weeks followed by avelumab once every 2 weeks plus M9241 once every 4 weeks at M9241 MTD until a criterion for treatment discontinuation has been met.
  Arms: Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg; Part B Cohort 1: UC Cohort Stage 1 combination therapy
Drug: M9241 (MTD) — Participants received M9241 at M9241 MTD once every 4 weeks until a criterion for treatment discontinuation has been met.
  Arms: Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg
Drug: Avelumab (Expansion cohort) — Participants in the expansion cohorts received Induction Therapy (Avelumab once weekly + M9241 once every 4 weeks) through Cycle 3 (for 12 weeks) then starting at Cycle 4, Continuation Therapy (Avelumab once every 2 weeks + M9241 once every 4 weeks).
  Arms: Part B Cohort 1: UC Cohort Stage 1 combination therapy

SUMMARY:
The study consisted of 2 parts: Dose Escalation phase (Part A) and Expansion phase (Part B). The dose escalation phase evaluated the safety, tolerability, and PK of avelumab in combination with M9241 in subjects with locally advanced, unresectable, or metastatic solid tumors. Expansion phase assessed the safety and clinical activity of the combination regimen in selected tumor types. In Expansion phase subjects who had completed the combination treatment of avelumab at a given dose level of M9241, a safety review was performed by the Safety monitoring committee in order to make a decision on the next dose level. Successive cohorts of 3 to 6 subjects were treated with escalating doses of M9241 with avelumab intravenous (IV).

ELIGIBILITY:
Inclusion Criteria:

Part A:

* subjects must had signed written informed consent.
* male or female subjects age greater than equals to (>=)18 years.
* subjects must had histologically or cytologically proven metastatic or locally advanced solid tumors for which no standard therapy exists, standard therapy had failed, subject was intolerant of established therapy known to provided clinical benefit for their condition, or standard therapy was not acceptable to subject.
* subjects who had been treated previously with a checkpoint inhibitor may enroll (except as outlined below for expansion cohorts).
* at least 1 unidimensional radiographically measurable lesion based on response evaluation criteria in solid tumors (recist) version 1. 1 (v1. 1), except for subjects with metastatic castration-resistant prostate cancer (crpc) or metastatic breast cancer who may been enrolled with objective evidence of disease without a measureable lesion. - eastern cooperative oncology group (ecog) performance status of 0 to 1 at screening
* estimated life expectancy of more than 12 weeks
* adequate hematological function as defined below:

  * white blood cells (wbc) count >= 3. 0 × 10^9 per liter (/l)
  * absolute neutrophil count >= 1. 5 × 10^9/l
  * lymphocyte count >= 0. 5 × 10^9/l
  * platelet count >= 100 × 10^9/l
  * hemoglobin >= 9 gram per deciliter (g/dl) (may had been transfused)
* adequate hepatic function as defined below:

  * a total bilirubin level less than equals to (<=) 1. 5 × upper limit of normal (uln) range
  * aspartate aminotransferase (ast) levels <= 2. 5 × uln (≤ 3 × uln for expansion cohorts)
  * alanine aminotransferase (alt) levels <= 2. 5 × uln (≤ 3 × uln for expansion cohorts)
  * subjects with documented gilbert disease were allowed if total bilirubin > 1. 5 but less than 3 × uln
* adequate renal function as defined by an estimated creatinine clearance >= 50 milliliter per minute (ml/min) according to cockcroft-gault formula
* negative blood pregnancy test at screening for women of childbearing potential. For purposes of this trial, women of childbearing potential were defined as all female subjects after puberty unless they were postmenopausal for at least 1 year, surgically sterile or sexually inactive.
* highly effective contraception (ie, methods with a failure rate of less than 1% per year) must been used before started of treatment, for duration of trial treatment, and for at least 50 days after stopping studied treatment for both men and women if risk of conception exists. The effects of avelumab and m9241 on developing human fetus were unknown; thus, women of childbearing potential and men agreed to use highly effective contraception.

Part B:

* Availability of a fresh tumor biopsy was mandatory for eligibility in the RCC cohort. The biopsy or surgical specimen should be collected within 28 days prior to the first IMP administration. If a subject had 2 separate biopsy attempts in which usable tissue was not obtained, enrollment would have been possible after discussion with the Medical Monitor. For other expansion cohorts, availability of either tumor archival material (< 6 months old) or fresh biopsies (obtained within 28 days) was acceptable with one of these being mandatory. For formalin-fixed paraffin-embedded samples, either block or sections (> 15) provided. Tumor biopsies and tumor archival material should have been suitable for biomarker assessment - Locally advanced or metastatic UC that had progressed during or after at least one previous platinum-based chemotherapy and not previously treated with anti-PD-1/PD-L1 agents: Histologically or cytologically confirmed locally advanced or metastatic transitional cell carcinoma of urothelium(including renal pelvis, ureters, urinary bladder, and urethra). Participants must had progressed during or after treatment with at least 1 platinum-containing regimen for inoperable locally advanced or metastatic UC or disease recurrence. Participants who had received prior adjuvant/neoadjuvant chemotherapy and progressed within 12 months of treatment with a platinum-containing regimen were considered as second line. Participants with mixed histologies were required to have a dominant transitional cell pattern.
* Non-small cell lung cancer (NSCLC), first-line metastatic: Stage IV (per seventh International Association for the Study of Lung Cancer classification) histologically confirmed NSCLC. Participants must not had received treatment for their metastatic disease. Participants could have received adjuvant chemotherapy or loco-regional treatment that included chemotherapy for locally advanced disease, as long as disease recurrence occurred at least 6 months after the completion of the last administration of chemotherapy. Only epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) wild-type were allowed (ie, EGFR mutation and ALK translocation / re arrangement excluded). Non squamous cell histologies and never / former light smoker (< 15 pack years) squamous cell carcinoma Participants (per local standard of care) required testing if status was unknown. Participants must had low tumor PD-L1 expression defined as < 50% tumor proportion score determined using PD-L1 IHC 22C3 pharmDx test or an equivalent Food and Drug Administration (FDA)- approved PD-L1 test. Availability of either tumor archival material or fresh biopsies within 28 days was acceptable with one of these being mandatory. For FFPE samples, either block or sections (> 15) may be provided. Tumor biopsies and tumor archival material had been suitable for biomarker assessment. This cohort would not be opened for enrollment in Belgium, Czech Republic, France, Germany, Hungary, Italy, Netherlands, Spain, and United Kingdom.
* Colorectal cancer (CRC): Histologically or cytologically confirmed recurrent or refractory metastatic CRC (according to American Joint Committee on Cancer / International Union Against Cancer Tumor Node Metastasis [TNM] Staging System seventh edition) after failure of prior therapy containing oxaliplatin / fluoropyrimidine and / or irinotecan / fluoropyrimidine and, if eligible, cetuximab (Erbitux®) and bevacizumab (Avastin®). Only Participants with microsatellite instability (MSI)-low or microsatellite stable (MSS) metastatic CRC are eligible. Participants without existing MSI test results had MSI status performed locally by a Clinical Laboratory Improvement Amendments (CLIA)-certified IHC or polymerase chain reaction (PCR)-based test (PCR based MSI test is preferred). Participants had to be willing to undergo an on-treatment biopsy procedure. Availability of either tumor archival material or fresh biopsies within 28 days was acceptable with one of these being mandatory. For FFPE samples, either a block or sections (> 15) could be provided. Tumor biopsies and tumor archival material had to be suitable for biomarker assessment. For Belgium, Czech Republic, France, Germany, Hungary, Italy, Netherlands, Spain, and United Kingdom, participants in the second-line setting had exhausted or were considered ineligible or intolerant (in the opinion of the Investigator) of available second-line chemotherapy options.
* Renal cell carcinoma (RCC), primary immune checkpoint inhibitor failure: Histologically or cytologically documented metastatic RCC with a component of clear cell subtype. Participants must have had progressive disease (PD) within 6 months or best overall response of stable disease (SD) for ≥ 6 months following start of therapy with any antibody / drug targeting T cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anticytotoxic T lymphocyte antigen-4 (CTLA-4) for advanced or metastatic disease (either as monotherapy or combination therapy, in any line). Fresh tumor biopsy was required for enrollment. If a subject had 2 separate biopsy attempts in which usable tissue was not obtained, enrollment could be possible after discussion with the Medical Monitor. Participants had to be willing to undergo an on-treatment biopsy procedure. In France, in addition to having received checkpoint inhibitor therapy, participants should have already received recommended local-standard therapy per discretion of the Investigator.

Exclusion Criteria:

* Concurrent treatment with a non-permitted drug/intervention (listed below)

  * Anticancer treatment (eg, cytoreductive therapy, radiotherapy, immune therapy, cytokine therapy, monoclonal antibody, targeted small molecule therapy) or any investigational drug within 4 weeks or 5 half-lives, whichever was shorter, prior to start of trial treatment, or not recovered from adverse event (AE) related to such therapies, with the following exceptions: Palliative radiotherapy delivered in a normal organ-sparing technique is permitted; Erythropoietin, darbepoetin-α and granulocyte colony-stimulating factor permitted; Hormonal therapies acting on the hypothalamic-pituitary-gonadal axis permitted (i.e. luteinizing hormone-releasing hormone agonist/antagonists). No other hormonal anticancer therapy was permitted.
  * Major surgery (as deemed by Investigator) for any reason, except diagnostic biopsy, within 4 weeks prior to start of trial treatment, or not fully recovered from surgery within 4 weeks prior to start of trial treatment.
  * Participants receiving immunosuppressive agents (such as steroids) for any reason were tapered off these drugs before start of trial treatment, with following exceptions: Participants with adrenal insufficiency, continued corticosteroids at physiologic replacement dose, equivalent to ≤ 10 mg prednisone daily; Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intra-ocular, or inhalation) was permitted; Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon was acceptable as long as it was anticipated that the administration of steroids would be completed in 14 days, or that the dose after 14 days would be equivalent to <= 10 mg prednisone daily.
* Any prior treatment with any form of interlukin-12 (IL-12)
* For the NSCLC, CRC, and UC expansion cohorts, prior therapy with any antibody / drug targeting T-cell co-regulatory proteins (immune checkpoints) such as anti-PD-1, anti-PD-L1, or anticytotoxic T lymphocyte antigen-4 (CTLA-4) antibody was prohibited.
* Intolerance to checkpoint inhibitor therapy, as defined by the occurrence of an AE requiring drug discontinuation. - Active or history of primary or metastatic central nervous system tumors
* Prior organ transplantation, including allogeneic stem-cell transplantation
* Previous malignant disease (other than the indication for this trial) within the last 5 years (except adequately treated non-melanoma skin cancers, carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least 2 years prior to trial entry and subject was deemed to have been cured with no additional therapy required or anticipated to be required.
* Significant acute or chronic infections requiring systemic therapy including, among others:

  • History of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome • Hepatitis B or C infection (HBV surface antigen positive and HBV core antibody positive with reflex to positive HBV deoxy ribonucleic acid (DNA) or HBV core antibody positive alone with reflex to positive HBV DNA or positive hepatitis C virus [HCV] antibody with reflex to positive HCV ribonucleic acid [RNA]). Participants with history of infection must had polymerase chain reaction documentation that infection was cleared.
* Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Participants with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment wer eligible if they wer stable on other medical treatment and do not fulfill exclusion criterion including Uncontrolled intercurrent illness - Known severe hypersensitivity reactions to monoclonal antibodies (Grade>= 3 National Cancer Institute-Common Terminology Criteria for Adverse Event (NCI-CTCAE) v4.03, or uncontrolled asthma (ie, 3 or more features of partially controlled asthma)
* History of allergic reaction to methotrexate (trace methotrexate may be present in M9241 as a part of manufacturing process) or history of severe hypersensitivity reaction to any other ingredient of study drug(s) and / or their excipients. Since M9241 contains sucrose as an excipient, participants suffering from hereditary fructose intolerance also excluded - Persisting toxicity related to prior therapy of Grade > 1 NCI-CTCAE v4.03 with the following exceptions:

  * Neuropathy Grade <= 2 was acceptable.
  * All grades of alopecia acceptable.
  * Endocrine dysfunction on replacement therapy was acceptable.
* Pregnancy or lactation
* Known alcohol or drug abuse as deemed by the Investigator
* Uncontrolled intercurrent illness including, but not limited to:

  * Hypertension uncontrolled by standard therapies (not stabilized to 150/90 millimeter of mercury (mm Hg) or lower)
  * Uncontrolled active infection
  * Uncontrolled diabetes (eg, glycosylated hemoglobin [HgbA1c] >= 8%)
* Clinically significant (or active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >= II), or serious cardiac arrhythmia requiring medication
* All other significant diseases (eg, inflammatory bowel disease, current severe acute or chronic colitis) or chronic medical conditions (including laboratory abnormalities) that in opinion of Investigator might impair subject's tolerance of trial treatment or interpretation of trial results.
* Any psychiatric condition that would prohibit understanding or endering of informed consent or that would limit compliance with trial requirements.
* Legal incapacity or limited legal capacity.
* Administration of a live vaccine within 30 days prior to trial entry.
* Any subject with possible area of ongoing necrosis (non-disease related), such as active ulcer, non-healing wound, or intercurrent bone fracture that may be at risk of delayed healing due to protocol therapy.
* Oxygen saturation < 90% at rest, known pulmonary fibrosis, or active interstitial lung disease.
* History of congenital or active immunodeficiency, with exception of acquired treatment-related hypogammaglobulinemia requiring periodic IV immunoglobulin infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (33):
- United States (17):
  - California Cancer Associates for Research & Excellence, Inc., San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Yale University Institutional Review Board, New Haven, Connecticut
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Hematology - Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Metairie Oncologists, LLC, Metairie, Louisiana
  - National Cancer Institute, Bethesda, Maryland
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - UC Health, LLC., Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cedar Sinai Medical Center, Ashland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Belgium (2):
  - Centre Hospitalier de l'Ardenne - Pharmacie, Libramont
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk
- France (6):
  - CHU Bordeaux - Hôpital Saint André, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital de la Timone# - CPCEM CIC - Bat F 1er étage, Marseille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Paul Strauss, Strasbourg
- Orszagos Onkologiai Intezet, Budapest, Hungary
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Netherlands (3):
  - Amsterdam UMC, Locatie VUMC, Amsterdam
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Hospital Universitario Virgen del Rocio, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- [Result] Strauss J, Deville JL, Sznol M, Ravaud A, Maruzzo M, Pachynski RK, Gourdin TS, Maio M, Dirix L, Schlom J, Donahue RN, Tsai YT, Wang X, Vugmeyster Y, Beier F, Seebeck J, Schroeder A, Chennoufi S, Gulley JL. First-in-human phase Ib trial of M9241 (NHS-IL12) plus avelumab in patients with advanced solid tumors, including dose expansion in patients with advanced urothelial carcinoma. J Immunother Cancer. 2023 May;11(5):e005813. doi: 10.1136/jitc-2022-005813. PMID 37236636
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201781_0031
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 parts: Part A (Dose escalation) and Part B (Dose expansion).
Pre-assignment Details: The study was conducted at 33 sites within Europe and the United States.
Groups:
- Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 4 micrograms per kilogram (mcg/kg) a subcutaneous (SC) injection at time (up to -20 minutes) relative to the start of Avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks on Day 1 and 15 during each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 12 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg (Experimental): Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg (Experimental): Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 800 milligrams (mg) IV infusion once weekly for the first 12 weeks, then 800 mg once every 2 weeks of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental): Participants in the expansion cohorts received M9241 at dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks on Day 1 in combination with Avelumab 800 mg IV infusion once weekly for the first 12 weeks, then 800 mg once every 2 weeks of each cycle (Each cycle=28 days) determined as the RP2D in the escalation part of the study.
Period: Overall Study
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg (Experimental) | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg (Experimental) | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Started | 9 | 7 | 7 | 6 | 7 | 16
Completed | 9 | 7 | 7 | 6 | 7 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg (Experimental) | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg (Experimental) | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental) | Total
Number analyzed (Participants) | 9 | 7 | 7 | 6 | 7 | 16 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 4 | 5 | 5 | 8 | 32
  >=65 years | 3 | 3 | 3 | 1 | 2 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 2 | 2 | 4 | 18
  Male | 4 | 5 | 4 | 4 | 5 | 12 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 6 | 7 | 6 | 5 | 16 | 48
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 1 | 0 | 3
  White | 7 | 5 | 6 | 6 | 6 | 8 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Event (NCI-CTCAE) v4.03
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs: reasonably related to the study intervention. Number of participants with TEAEs and treatment related TEAEs were reported.
Time Frame: From first dose of study treatment up to 1311 days
Population: Safety analysis set (SAF) included all participants who receive at least 1 dose (complete or incomplete) of any investigational medicinal product (IMP) (Avelumab or NHS-IL12).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6 | 7
Participants
  Participants with TEAEs | 9 | 7 | 7 | 6 | 7
  Participants with Treatment-related-TEAEs | 8 | 5 | 6 | 5 | 6

2. Primary Outcome: Part B: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Event (NCI-CTCAE) v4.03
Description: as for outcome 1
Time Frame: Part B: From first dose of study treatment up to 443 days
Population: SAF included all participants who receive at least 1 dose of any investigational medicinal product (IMP) (Avelumab or NHS-IL12).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
Participants
  Participants with TEAEs | 16
  Participants with Treatment-Related AEs | 15

3. Primary Outcome: Part A: Number of Participants With Treatment-Related Adverse Events (TRAEs) by Severity Based on Grade 3,4 and 5 According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: AE was any untoward medical occurrence in a participants who received study drug without regard to possibility of causal relationship. An AE was considered treatment emergent if occurred for the first time after the start of study treatment or occurred prior to the start of treatment. Severity of TEAEs were graded using NCI-CTCAE v4.03 toxicity grades, as follows: Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with Grade 3,4 and 5 by severity were only reported.
Time Frame: From first dose of study treatment up to 1311 days
Population: SAF analysis set included all participants who receive at least 1 dose (complete or incomplete) of any IMP (Avelumab or NHS-IL12).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6 | 7
Participants
  Grade >=3 | 6 | 5 | 6 | 4 | 4
  Grade >=4 | 2 | 2 | 2 | 2 | 1
  Grade 5 | 0 | 1 | 0 | 1 | 1

4. Primary Outcome: Part B: Number of Participants With Treatment-Related Adverse Events (TRAEs) by Severity According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: AE was any untoward medical occurrence in a participants who received study drug without regard to possibility of causal relationship. An AE was considered treatment emergent if occurred for the first time after the start of study treatment or occurred prior to the start of treatment. Severity of TEAEs were graded using NCI-CTCAE v4.03 toxicity grades, as follows: Grade 1= Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with TEAEs and TRAEs by severity were reported.
Time Frame: First dose of study drug up to 443 days
Population: SAF analysis set included all participants who receive at least 1 dose (complete or incomplete) of any IMP (Avelumab or NHS-IL12). Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 15
Participants
  Any Grade | 15
  Grade >=3 | 8
  Grade >=4 | 1
  Grade 5 | 0

5. Primary Outcome: Part A: Number of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: A DLT is any Grade (>=) 3 non-hematologic AE or any Grade (>=) 4 hematologic AE according to the NCI-CTCAE v4.03, occurring during the DLT observation period that is related to either or both study drugs as determined by the Investigator or Sponsor at any dose and judged not to be related to the underlying disease or any previous or concomitant medication. The following are exceptions to the DLTs: Grade >=3 thrombocytopenia with medically concerning bleeding; Any Grade 3 autoimmune thyroid-related toxicity that doesn't clinically resolve to <= Grade 2 within 7 days of initiating therapy will be a DLT. Any Grade 4 neutropenia of < 5 days duration; Grade 3 infusion-related reaction resolving within 6 hours of infusion; Grade 3 diarrhea or skin toxicity that resolves to Grade <= 1 within 7 days after medical management; Transient Grade 3 fatigue, local reactions, flu-like symptoms; Tumor flare phenomenon of known or suspected tumor did not consider a DLT.
Time Frame: Time from first treatment to final assessment up to 3 weeks
Population: DLTs analysis set included all participants who received all treatment in the DLT period or stopped treatment because of DLTs in the DLT period.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg: Participants received M9241 at a dose of 8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 7
Participants | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Part B: Number of Participants With Confirmed Best Overall Response (BOR) Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Confirmed BOR was defined as the best response of any of the confirmed complete response (CR), confirmed partial response (PR), stable disease (SD) and progressive disease (PD) recorded from the date of randomization until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference).CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)= Neither sufficient increase to qualify for progression of disease (PD) nor sufficient shrinkage to qualify for PR. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Not evaluable (NE): No post-baseline assessment. BOR assessments were assessed by investigators.
Time Frame: First dose of study drug up to 443 days
Population: Full analysis set included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 2
  Progressive Disease | 13
  Not evaluable | 1

7. Secondary Outcome: Part A: Area Under Serum Concentration Time Curve From Time Zero to the Time of the Last Observation (AUC0-t) of Avelumab
Description: Area under the serum concentration versus time curve from time zero to the last sampling time t at which concentration is at or above the lower limit of quantification (LLLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Predose (PrD),1,4,8 hours postdose (PD) on Day 1,22 of Cycle 1 & 2; PrD,1 hour PD on Day 8,15 of Cycle 1 & Day 8,15,22 of Cycle 2; PrD, 1 hour PD on Day 1 Cycle 3 & Day 1,15 of Cycle 4; PrD on Day 1 of Cycle 7,10,13,16,19,22,25, & 28 (Each cycle: 28 days)
Population: Pharmacokinetic analysis set included all participants who completed at least 1 administration of avelumab and/or M9241, and who provided at least 1 sample with a measurable concentration of avelumab or M9241. Here, "Overall Number of participants analyzed", signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
microgram*hour per milliliter (mcg*h/mL)
  Cycle 1 Day 1 | 20700 (38.1) | 26600 (57.9) | 23600 (16.6) | 17400 (33.4) | 17900 (39.7)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5 | 5 | 6 | 0
  Cycle 1 Day 15 | 22800 (40.5) | 26100 (42.5) | 28300 (39.4) | 22000 (19.2) |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5
  Cycle 1 Day 22 |  |  |  |  | 26300 (31.0)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 5 | 7
  Cycle 2 Day 1 | 26400 (17.2) | 27900 (47.9) | 22700 (23.2) | 22700 (10.5) | 22100 (42.7)
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Part A: Area Under Serum Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Avelumab
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: PrD, 1, 4, 8 hours PD on Day 1, 22 of cycle 1 & 2; PrD, 1 hour PD on Day 8, 15 of cycle 1 & Day 8, 15, 22 of cycle 2; PrD, 1 hour PD on Day 1 cycle 3 & Day 1, 15 of cycle 4; PrD on Day 1 of cycle 7, 10,13,16,19,22,25, & 28 (Each cycle: 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
microgram*hour per milliliter (mcg*h/mL)
  Cycle 1 Day 1 | 22300 (41.5) | 30100 (75.8) | 26500 (21.5) | 18800 (29.5) | 27000 (65.0)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 5 | 5 | 4 | 0
  Cycle 1 Day 15 | 26300 (37.2) | 29800 (35.7) | 27100 (34.5) | 23000 (26.0) |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 22 |  |  |  |  | 43400 (56.1)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 4 | 7
  Cycle 2 Day 1 | 29800 (18.4) | 33100 (48.4) | 24300 (30.6) | 24400 (13.3) | 35100 (40.3)
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part A: Terminal Elimination Rate Constant (Lambdaz) of Avelumab
Description: Lambda(z) was determined from the terminal slope of the log-transformed serum concentration curve using linear regression method.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: One per hour (1/hour)
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
One per hour (1/hour)
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 7 | 7 | 6 | 6
  Cycle 1 Day 1 | 0.00847 (29.6) | 0.00729 (48.5) | 0.00756 (20.6) | 0.00790 (14.4) | 0.00822 (37.1)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 5 | 4 | 4 | 0
  Cycle 1 Day 15 | 0.00780 (31.6) | 0.00814 (15.7) | 0.00780 (31.4) | 0.00803 (17.1) |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 22 |  |  |  |  | 0.00620 (34.3)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 4 | 4 | 7
  Cycle 2 Day 1 | 0.00659 (15.7) | 0.00714 (39.8) | 0.00868 (19.2) | 0.00830 (16.4) | 0.00793 (35.9)
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Part A: Maximum Observed Serum Concentration (Cmax) of Avelumab
Description: Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
microgram/milliliter (mcg/mL)
  Cycle 1 Day 1 | 241 (39.9) | 244 (29.9) | 287 (36.4) | 156 (67.7) | 228 (29.3)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5 | 4 | 4 | 0
  Cycle 1 Day 15 | 229 (54.4) | 250 (14.6) | 256 (32.0) | 201 (25.6) |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5
  Cycle 1 Day 22 |  |  |  |  | 269 (44.0)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 4 | 7
  Cycle 2 Day 1 | 213 (21.3) | 249 (37.5) | 210 (19.7) | 200 (8.1) | 318 (33.5)
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part A: Minimum Observed Serum Concentration (Cmin) of Avelumab
Description: Cmin is minimum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg: Participants received M9241 at a dose of 4 micrograms per kilogram (mcg/kg) a subcutaneous (SC) injection at time (up to -20 minutes) relative to the start of Avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks on Day 1 and 15 during each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 7
mcg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5 | 5 | 6 | 0
  Cycle 1 Day 15 | 11.3 (90.4) | 14.5 (37.2) | 14.0 (70.3) | 9.28 (51.8) |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5
  Cycle 1 Day 22 |  |  |  |  | 74.1 (62.0)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 5 | 7
  Cycle 2 Day 1 | 20.5 (37.6) | 24.0 (79.9) | 14.4 (91.9) | 13.1 (24.4) | 59.3 (122.5)
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part A: Time to Reach Maximum Observed Concentration (Tmax) of Avelumab
Description: Tmax is time to reach maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Groups:
- Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg: Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
hours
  Cycle 1 Day 1 | 4.00 [1.00 to 25.08] | 1.05 [1.00 to 9.00] | 3.90 [1.00 to 4.25] | 2.58 [1.00 to 44.78] | 4.00 [1.00 to 22.20]
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5 | 4 | 4 | 0
  Cycle 1 Day 15 | 5.04 [1.00 to 48.42] | 1.13 [1.00 to 25.72] | 4.00 [1.22 to 49.00] | 4.09 [1.03 to 29.18] |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5
  Cycle 1 Day 22 |  |  |  |  | 4.00 [1.00 to 43.03]
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 4 | 7
  Cycle 2 Day 1 | 1.58 [1.13 to 25.00] | 1.17 [1.10 to 4.08] | 23.07 [3.98 to 25.00] | 2.00 [1.00 to 25.35] | 4.00 [1.12 to 9.00]
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Part A: Apparent Terminal Half-life (t1/2) of Avelumab
Description: Apparent terminal half-life was defined as the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
hours
  Cycle 1 Day 1 | 94.7 [48.4 to 108] | 87.4 [50.2 to 223] | 95.2 [70.1 to 123] | 87.1 [69.4 to 106] | 70.5 [60.2 to 148]
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5 | 4 | 4 | 0
  Cycle 1 Day 15 | 101 [54.9 to 115] | 77.6 [75.0 to 103] | 84.1 [65.0 to 136] | 86.7 [69.9 to 106] |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5
  Cycle 1 Day 22 |  |  |  |  | 102 [83.3 to 180]
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 4 | 4 | 7
  Cycle 2 Day 1 | 106 [88.5 to 125] | 94.9 [68.6 to 173] | 80.7 [67.5 to 95.1] | 86.2 [67.0 to 98.1] | 81.1 [55.9 to 138]
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Part A: Area Under the Serum Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of Avelumab
Description: AUCtau was defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Groups:
- Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg; Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg: Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 800 milligrams (mg) IV infusion once weekly for the first 12 weeks, then 800 mg once every 2 weeks of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 8 | 7 | 7 | 6 | 7
mcg*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 8 | 7 | 7 | 6 | 6
  Cycle 1 Day 1 | 20900 (37.6) | 26700 (58.3) | 24500 (19.2) | 17400 (33.1) | 19800 (44.7)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 5 | 4 | 4 | 0
  Cycle 1 Day 15 | 24100 (35.0) | 27600 (33.1) | 28300 (39.4) | 21400 (24.2) |
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
  Cycle 1 Day 22 |  |  |  |  | 27500 (34.7)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 4 | 7
  Cycle 2 Day 1 | 26400 (17.4) | 29500 (37.6) | 22900 (27.1) | 22800 (11.6) | 25500 (26.1)
  Cycle 2 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Part A: Area Under Serum Concentration Time Curve From Time Zero to the Time of the Last Observation (AUC0-t) of M9241
Description: Area under the serum concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the lower limit of quantification (LLLQ). (AUC0-t) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: PrD, 1, 4, 8 hours PD on Day 1 of cycle 1 and Day 1 of cycle 2; PrD on Day 15 of cycle 1 and cycle 2; PrD, 1hour PD on Day 1 of cycle 3 and cycle 4; PrD on Day 1 Cycle 7, 10, 13, 16, 19, 22, 25, and 28 (Each cycle: 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 7
nanogram*hour/milliliter (ng*h/mL)
  Cycle 1 Day 1 | 105 (114.4) | 421 (82.9) | 661 (58.2) | 621 (96.5) | 873 (264.0)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 5 | 7
  Cycle 2 Day 1 | 183 (151.7) | 306 (132.6) | 184 (174.0) | 1250 (46.2) | 1060 (308.8)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Part A: Area Under Serum Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M9241
Description: as for outcome 8
Time Frame: as for outcome 15
Population: Pharmacokinetic analysis set included participants who completed at least 1 administration of avelumab and/or M9241 and provided at least 1 sample with a measurable concentration. Here, "Overall Number of participants analyzed", signifies participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable at the specified time point. None of the participants were analyzed in Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg arm at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg: Participants received subcutaneous (SC) injection of M9241 at a dose of 4 micrograms per kilogram (mcg/kg) once every 4 week on Day 1 in combination with IV infusion of Avelumab 10 milligrams per kg (mg/kg) once every 2 weeks on Day 1 and 15 of each cycle (each cycle is of 28 days) until any criterion for treatment discontinuation were met
- Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg: Participants received SC injection of M9241 at a dose of 8 mcg/kg once every 4 week on Day 1 in combination with IV infusion of Avelumab 10 mg/kg once every 2 weeks on Day 1 and 15 of each cycle (each cycle is of 28 days) until any criterion for treatment discontinuation were met
- Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg: Participants received SC injection of M9241 at a dose of 12 mcg/kg once every 4 week on Day 1 in combination with IV infusion of Avelumab 10 mg/kg once every 2 weeks on Day 1 and 15 of each cycle (each cycle is of 28 days) until any criterion for treatment discontinuation were met
- Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg: Participants received IV infusion of avelumab at dose of 800 mg once weekly for the first 12 weeks in combination with SC injection of M9241, 16.8 mcg/kg once every 4 weeks, then avelumab at 800 mg IV infusion once every 2 weeks in combination with M9241 at dose of 16.8 mcg/kg SC injection once every 4 weeks until criteria for treatment discontinuation were met
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 0 | 2 | 1 | 2 | 4
ng*h/mL
  Cycle 1 Day 1 |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 2370 (31.5)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3
  Cycle 2 Day 1 |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 2860 (19.9)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part A: Terminal Elimination Rate Constant (Lambdaz) of M9241
Description: as for outcome 9
Time Frame: PrD, 1, 4, 8 hours PD on Day 1 of cycle 1 and Day 1 of cycle 2; PrD on Day 15 of cycle 1 and cycle 2; PrD, 1 hour PD on Day 1 of cycle 3 and cycle 4; PrD on Day 1 Cycle 7, 10, 13, 16, 19, 22, 25, and 28 (Each cycle: 28 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: One per hour (1/hour)
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 0 | 2 | 1 | 2 | 4
One per hour (1/hour)
  Cycle 1 Day 1 |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 0.00451 (12.5)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3
  Cycle 2 Day 1 |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 0.00835 (14.0)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Part A: Maximum Observed Serum Concentration (Cmax) of M9241
Description: Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 7
ng/mL
  Cycle 1 Day 1 | 2.79 (79.1) | 4.42 (84.9) | 12.6 (40.9) | 5.91 (54.8) | 6.88 (99.6)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 5 | 7
  Cycle 2 Day 1 | 2.68 (45.7) | 3.81 (39.4) | 4.45 (112.8) | 9.42 (63.3) | 10.4 (134.1)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Part A: Minimum Observed Serum Concentration (Cmin) of M9241
Description: Cmin is minimum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 7
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Part A: Time to Reach Maximum Observed Concentration (Tmax) of M9241
Description: Tmax is time to reach maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 7
hours
  Cycle 1 Day 1 | 25.08 [24.58 to 26.05] | 25.17 [3.17 to 240.73] | 24.11 [9.02 to 42.73] | 36.17 [9.17 to 238.62] | 25.08 [19.03 to 46.40]
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 5 | 5 | 5 | 7
  Cycle 2 Day 1 | 34.28 [9.33 to 44.45] | 25.17 [10.13 to 45.03] | 25.08 [9.27 to 47.88] | 25.43 [10.10 to 94.93] | 25.50 [9.35 to 168.18]
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
  Cycle 4 Day 1 |  |  |  |  | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 00
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Part A: Apparent Terminal Half-life (t1/2) of M9241
Description: as for outcome 13
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 0 | 2 | 1 | 2 | 4
hours
  Cycle 1 Day 1 |  | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 161 [128 to 169]
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3
  Cycle 2 Day 1 |  | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. |  | NA [NA to NA] — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 84.4 [71.6 to 94.6]
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Part A: Area Under the Serum Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of M9241
Description: as for outcome 14
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 0 | 2 | 2 | 5 | 5
ng*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 2 | 2 | 5 | 4
  Cycle 1 Day 1 |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 835 (64.3) | 2130 (35.6)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 2 | 5
  Cycle 2 Day 1 |  | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values. | 2390 (80.4)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Part A: Number of Participants With At Least One Positive Anti-drug Antibodies (ADA) for Avelumab and M9241
Description: ADA category of each participant was classified as pre-existing immunoreactivity (positive ADA response at baseline (prior to treatment), treatment-boosted (positive response at baseline with at least one post baseline titer at >=8-fold baseline titer), or treatment-emergent (TE [any positive post baseline assay response when baseline results were negative or missing or not reported]). TE ADA responses were further classified as persistent (treatment-emergent positive ADA response detected in at least 2 consecutive post baseline samples separated by at least a 16-week post baseline period [based on nominal sampling time], with no ADA-negative samples in-between or positive response at last ADA sampling time point) and transient (not persistent/indeterminate, regardless of any missing samples).
Time Frame: First dose of study drug up to 1311 days
Population: Immunogenicity analysis set included all participants who received at least 1 complete dose (at least 90% of planned dose) of any study treatment & at least 1 valid ADA result for avelumab or NHS-IL12.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6 | 7
Participants
  Avelumab: ADA pre-existing | 0 | 0 | 0 | 0 | 1
  Avelumab: ADA Treatment boosted | 0 | 0 | 0 | 0 | 0
  Avelumab: Treatment-Emergent Transient positive | 0 | 0 | 1 | 1 | 0
  Avelumab: Treatment-Emergent Persistent Positive | 0 | 1 | 1 | 0 | 1
  M9241: ADA pre-existing | 0 | 0 | 0 | 0 | 0
  M9241: ADA Treatment boosted | 0 | 0 | 0 | 0 | 0
  M9241: Treatment-Emergent Transient Positive | 0 | 0 | 0 | 0 | 0
  M9241: Treatment-Emergent Persistent Positive | 0 | 0 | 0 | 0 | 1

24. Secondary Outcome: Part A: Number of Participants With Confirmed Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1
Description: BOR is defined as best response of any of confirmed complete response, confirmed partial response, stable disease and progressive disease recorded from date of randomization until disease progression or recurrence. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)= Neither sufficient increase to qualify for progression of disease (PD) nor sufficient shrinkage to qualify for PR. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. Non-CR/non-PD (for participants with non-measurable disease at baseline) = at least one Non-CR/non-PD assessment (or better) >= 6 weeks after first study treatment administration and before progression and Not Evaluable: all other cases. BOR assessments were assessed by investigators.
Time Frame: First dose of study drug up to 1311 days
Population: Full analysis set included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6 | 7
Participants
  Complete Response (CR) | 0 | 1 | 0 | 1 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 2 | 2 | 2 | 1 | 2
  Progressive Disease (PD) | 6 | 3 | 4 | 2 | 5
  Non CR/Non PD | 0 | 0 | 0 | 0 | 0
  Not Evaluable | 1 | 1 | 1 | 2 | 0

25. Secondary Outcome: Pat A: Number of Participants With Immune-related Best Overall Response (BOR) Using Immune-related Response Criteria Derived From Response Evaluation Criteria in Solid Tumors Version 1.1
Description: BOR: best response of any of immune related complete response (irCR), immune related partial response (irPR), immune related stable disease (irSD) and immune related progressive disease (irPD) recorded from the date of randomization until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). irCR: Complete disappearance of all tumor lesions (both index and non-index lesions with no new measurable/unmeasurable lesions). irPR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions). irSD: SLD of target and new measurable lesions neither irCR, irPR, or irPD. irPD: SLD of target and new measurable lesions increases greater than or equal to [>=] 20%, confirmed by a repeat, consecutive observations at least 4 weeks from the date first documented. Number of participants with immune-related best overall response in each category (irCR, irPR, irSD, irPD) was reported.
Time Frame: First dose of study drug up to 1311 days
Population: Full analysis set included all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 2: M9241 8 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg + Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg + Avelumab 800 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6 | 7
Participants
  Immune-Related Complete Response (irCR) | 0 | 1 | 0 | 1 | 0
  Immune-Related Partial Response (irPR) | 0 | 0 | 0 | 0 | 0
  Immune-Related Stable Disease (irSD) | 2 | 2 | 2 | 3 | 3
  Immune-Related Progressive Disease (irPD) | 0 | 0 | 0 | 0 | 2
  Not evaluable (NE) | 7 | 4 | 5 | 2 | 2

26. Secondary Outcome: Part B: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Criteria Assessed by Investigator
Description: PFS was defined as the time from first treatment day until date of the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier estimates.
Time Frame: Time from first dose administration until progressive disease or death, assessed up to 443 days
Population: Full analysis set included all participants who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
weeks | 7.6 (7.1) [7.1 to 8.0]

27. Secondary Outcome: Part B: Overall Survival (OS) Time
Description: The OS time was defined as the time from treatment day 1 to the date of death due to any cause. The participants who were still alive at the time of data analysis or who were lost to follow-up OS time was censored at the last recorded date that the participant was known to be alive before the data cutoff date. OS was measured using Kaplan-Meier estimates.
Time Frame: Time from first dose of study treatment up to 443 days
Population: Full analysis set included all participants who received at least 1 dose of any study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
months | 4.9 (2.3) [2.3 to 11.8]

28. Secondary Outcome: Part B: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Criteria Assessed by Investigator
Description: DOR according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and as assessed by an Investigator was defined as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of objective progression of disease (PD) or death due to any cause whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. If a participant has not an event (PD or death), DOR was censored at the date of last adequate tumor assessment.
Time Frame: Time from first dose of study treatment up to 443 days
Population: Data could not be calculated as none of the participants showed objective response.
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 0

29. Secondary Outcome: Part B: Maximum Observed Serum Concentration (Cmax) of M9241
Description: Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 1 hour post-dose on Day 1 and Day 29 of Cycle 1 and 2 (Each cycle: 28 days)
Population: Pharmacokinetic analysis set included all participants who completed at least 1 administration of avelumab and/or M9241, and who provided at least 1 sample with a measurable concentration of avelumab or M9241. Here "Number analyzed" signifies those participants who were evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
ng/mL
  Day 1 | 6.95 (59.6)
  Day 29: number analyzed (Participants) | 11
  Day 29 | 7.62 (113.0)

30. Secondary Outcome: Part B: Serum Trough Concentration Levels (Ctrough) of M9241
Description: Ctrough was defined as the trough or minimum serum concentration.
Time Frame: Pre-dose, 1 hour post-dose on Day 1 of cycle 2; Day 1, 27 of cycle 3; Day 1 of cycle 5 (Each cycle: 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 12
ng/mL
  Day 29 | 0 (0)
  Day 57: number analyzed (Participants) | 5
  Day 57 | 0 (0)
  Day 83: number analyzed (Participants) | 2
  Day 83 | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.
  Day 113: number analyzed (Participants) | 2
  Day 113 | NA (NA) — Based on pre-specified criteria, statistical analysis for PK was only performed if more than 3 participants have reportable parameter values.

31. Secondary Outcome: Part B: Concentration at the End of Infusion (Ceoi) of Avelumab
Description: Ceoi is the observed serum drug concentration at the end of Intravenous (IV) infusion.
Time Frame: Pre-dose, 1 hour post-dose on Day 1 and 15 of Cycle 1 and 2 (Each cycle: 28 days)
Population: Pharmacokinetic analysis set included all participants who completed at least 1 administration of avelumab and/or M9241, and who provided at least 1 sample with a measurable concentration of avelumab or M9241. Here, "Number analyzed" signifies those participants who were evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
mcg/mL
  Day 1 | 199 (22.0)
  Day 15: number analyzed (Participants) | 11
  Day 15 | 220 (37.9)
  Day 29: number analyzed (Participants) | 12
  Day 29 | 272 (59.6)
  Day 43: number analyzed (Participants) | 12
  Day 43 | 253 (40.0)

32. Secondary Outcome: Part B: Serum Trough Concentration Levels (Ctrough) of Avelumab
Description: Ctrough was defined as the trough or minimum serum concentration.
Time Frame: Pre-dose, 1 hour post-dose on Day 15, 29 and 43
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 13
mcg/mL
  Day 15 | 54.2 (64.9)
  Day 29: number analyzed (Participants) | 12
  Day 29 | 53.9 (217.5)
  Day 43: number analyzed (Participants) | 12
  Day 43 | 44.6 (101.8)

33. Secondary Outcome: Part B: Number of Participants With At Least One Positive Anti-drug Antibodies (ADA) of Avelumab and M9241
Description: as for outcome 23
Time Frame: Time from first dose of study treatment up to 443 days
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
Number analyzed (Participants) | 16
Participants
  Avelumab: ADA pre-existing | 0
  Avelumab: ADA treatment boosted | 0
  Avelumab: Treatment-Emergent Transient Positive | 0
  Avelumab: Treatment-Emergent Persistent Positive | 1
  M9241: ADA pre-existing | 0
  M9241: ADA treatment boosted | 0
  M9241: Treatment-Emergent Transient Positive | 1
  M9241: Treatment-Emergent Persistent Positive | 0

ADVERSE EVENTS:
Time Frame: Part A: Baseline up to 1311 days Part B: Baseline up to 443 days
Groups:
- Part A Cohort 2: M9241 8 mcg/kg +Avelumab 10 mg/kg: Participants received M9241 at a dose of 8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part A Cohort 3: M9241 12 mcg/kg +Avelumab 10 mg/kg: Participants received M9241 at a dose of 12 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 10 mg/kg IV infusion every 2 weeks on Day 1 and 15 of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
- Part A Cohort 5: M9241 16.8 mcg/kg +Avelumab 800 mg: Participants received M9241 at a dose of 16.8 mcg/kg SC injection at time (up to -20 minutes) relative to the start of avelumab infusion (time 0), once every 4 weeks, on Day 1 in combination with Avelumab 800 milligrams (mg) IV infusion once weekly for the first 12 weeks, then 800 mg once every 2 weeks of each cycle (Each cycle=28 days) until any criterion for treatment discontinuation were met.
Arm/Group | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental) | Part A Cohort 2: M9241 8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 3: M9241 12 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg | Part A Cohort 5: M9241 16.8 mcg/kg +Avelumab 800 mg | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental)
All-Cause Mortality (participants affected / at risk) | 9/9 | 5/7 | 6/7 | 5/6 | 7/7 | 12/16
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/7 | 3/7 | 3/6 | 4/7 | 12/16
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7 | 7/7 | 6/6 | 7/7 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental) (N=9) | Part A Cohort 2: M9241 8 mcg/kg +Avelumab 10 mg/kg (N=7) | Part A Cohort 3: M9241 12 mcg/kg +Avelumab 10 mg/kg (N=7) | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg (N=6) | Part A Cohort 5: M9241 16.8 mcg/kg +Avelumab 800 mg (N=7) | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental) (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 1 | 1 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: M9241 4 mcg/kg + Avelumab 10 mg/kg (Experimental) (N=9) | Part A Cohort 2: M9241 8 mcg/kg +Avelumab 10 mg/kg (N=7) | Part A Cohort 3: M9241 12 mcg/kg +Avelumab 10 mg/kg (N=7) | Part A Cohort 4: M9241 16.8 mcg/kg +Avelumab 10 mg/kg (N=6) | Part A Cohort 5: M9241 16.8 mcg/kg +Avelumab 800 mg (N=7) | Part B Cohort 1: UC Cohort Stage 1 Combination Therapy (Experimental) (N=16)
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 5 | 4 | 3 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 1 | 1 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 4 | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 2 | 6
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 3 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 4 | 0 | 2 | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 5 | 3 | 4 | 4 | 10
Fatigue (General disorders) | 7 | 3 | 4 | 2 | 4 | 0
Influenza like illness (General disorders) | 4 | 4 | 2 | 3 | 0 | 0
Chills (General disorders) | 2 | 2 | 1 | 2 | 2 | 6
Oedema peripheral (General disorders) | 4 | 1 | 0 | 0 | 0 | 3
Malaise (General disorders) | 0 | 1 | 1 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 7
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 4
Injection site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 2 | 0 | 2 | 3
Alanine aminotransferase increased (Investigations) | 2 | 1 | 2 | 1 | 1 | 4
Lymphocyte count decreased (Investigations) | 4 | 4 | 3 | 4 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 3 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 1 | 0 | 1 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2
Weight increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3 | 4 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 3
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 1 | 1 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 (0) | 1 (1) | 0 | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 2 | 3 | 1
Headache (Nervous system disorders) | 1 | 3 | 0 | 1 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Resting tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 3 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 3 | 0 | 1 | 3 | 0 | 2
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 0 | 1 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hydroureter (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary fistula (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to pre-specified futility criteria met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT02994953/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT02994953/SAP_001.pdf